CLINICAL TRIAL: NCT00344422
Title: A Multi-Center Randomized Study of Vincristine, Doxil and Dexamethasone vs. Vincristine, Doxorubicin, and Dexamethasone in Patients With Multiple Myeloma
Brief Title: Vincristine, DOXIL (Doxorubicin HCl Liposome Injection) and Dexamethasone vs. Vincristine, Doxorubicin, and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002434
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Multiple Myeloma; Myeloma; M-Protein; Myeloma Proteins
Keywords: Anthracyclines; Liposomes; Liposomal; Vincristine; Doxorubicin; Dexamethasone; Pegylated Liposomal Doxorubicin; DOXIL; drug resistant myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Vincristine; liposomal doxorubicin; Dexamethasone; Doxorubicin

INTERVENTIONS:
Drug: Vincristine, DOXIL (doxorubicin HCl liposomal injection), and Dexamethasone (VDD) vs. Vincristine, Doxorubicin and Dexamethasone (VAD)

SUMMARY:
The purpose of this study is to determine how well newly diagnosed multiple myeloma patients respond to an experimental regimen of Vincristine, DOXIL (doxorubicin HCl liposome injection) and Dexamethasone (VDD) versus the standard treatment of Vincristine, Doxorubicin and Dexamethasone (VAD).

DETAILED DESCRIPTION:
This is a randomized, open label study comparing the efficacy, clinical benefit, toxicity and safety of the combination of Vincristine, DOXIL® (doxorubicin HCl liposome injection), and Dexamethasone (VDD) to the standard regimen of Vincristine, Doxorubicin and Dexamethasone (VAD) in patients with newly diagnosed multiple myeloma. Approximately 200 patients with newly diagnosed multiple myeloma will be randomized to receive either VDD or VAD. This study will determine and compare the objective response rate (the percentage of patients who attain an Objective Status of Complete Remission, Remission or Partial Remission) for patients receiving VDD vs. VAD. This study will also evaluate and compare the clinical benefit of VDD vs. VAD for the following measures: Hospitalization; Documented sepsis; Antibiotic use; Grade 3 or 4 neutropenia or neutropenic fever.

VDD: Vincristine 1.4 mg/m2 IV on Day 1; Doxil® 40 mg/m2 IV on Day 1; Dexamethasone 40 mg/day oral Days 1-4; VAD: Vincristine 0.4 mg/day continuous infusion Days 1-4; Doxorubicin 9.0 mg/m2/day continuous infusion Days 1-4; Dexamethasone 40 mg/day orally on Days 1-4; Every 28 days for 4 cycles

ELIGIBILITY:
Inclusion Criteria:

* Untreated multiple myeloma requiring treatment
* Total cumulative dose of prior doxorubicin can not exceed 240 mg/m2
* Must have measurable disease
* Left Ventricular Ejection Fraction (LVEF) >= 50 % determined by Multiple Gated Acquisition Scan (MUGA)
* Karnofsky performance status of >= 60%
* Adequate bone marrow, liver and renal function
* Disease-free from prior malignancies >= 5 years with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Female participants (if of child bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) must use medically acceptable methods of birth control.

Exclusion Criteria:

* Life expectancy of >= 3 months
* Pregnant or breast feeding
* History of cardiac disease, with New York Heart Association Class II or greater, with congestive heart failure
* or unstable angina, uncontrolled hypertension or cardiac arrythmias or myocardial infarction within the last 6 months
* Uncontrolled diabetes mellitus or systemic infection
* Nonsecretory myeloma, Monoclonal Gammopathy of Unknown Significance (MGUS) or smoldering myeloma
* Confusion, disorientation, or history of psychiatric illness which may impair patient's ability to give informed consent
* Prior chemotherapy to treat Multiple Myeloma
* Prior radiotherapy to an area greater than 1/3 of the skeleton
* Prior local radiotherapy within 1 week of treatment
* Any investigational agent within 30 days of the first dose of treatment
* Prior single agent dexamethasone (or another corticosteroid) to treat Multiple Myeloma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2000-10; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
To determine and compare the objective response rate (the percentage of patients who attain an Objective Status of Complete Remission, Remission or Partial Remission) for patients receiving VDD vs VAD.

SECONDARY OUTCOMES:
To evaluate and compare the clinical benefit of VDD vs VAD for the following measures: Hospitalization, Documented sepsis,Antibiotic use, Grade 3 or 4 neutropenia or neutropenic fever

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Rifkin RM, Gregory SA, Mohrbacher A, Hussein MA. Pegylated liposomal doxorubicin, vincristine, and dexamethasone provide significant reduction in toxicity compared with doxorubicin, vincristine, and dexamethasone in patients with newly diagnosed multiple myeloma: a Phase III multicenter randomized trial. Cancer. 2006 Feb 15;106(4):848-58. doi: 10.1002/cncr.21662. PMID 16404741
- See also: A Multi-Center Randomized Study of Vincristine, DOXIL and Dexamethasone vs. Vincristine Doxorubicin, and Dexamethasone in Patients with Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=479&filename=CR002434_CSR.pdf